CLINICAL TRIAL: NCT04293874
Title: Association Between Dietary Omega-3 Fatty Acid Intake Patterns and Psychoneurological Symptoms in Women Following Treatment for Early-stage Breast Cancer
Brief Title: Adaptive Symptom Care Using Fish-Based Nutritional Directives Post Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Collaborators: Hartford HealthCare (Other); Seafood Industry Research Fund (Unknown); Alaskan Seafood Marketing Institute (Unknown); Academy of Nutrition and Dietetics (Other)
Responsible Party: Principal Investigator, Michelle Judge, Associate Professor, University of Connecticut
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-HHC-2016-0245
Record Dates: First submitted 2020-02-27; First posted 2020-03-03 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Fatigue; Depression; Pain; Sleep Disturbance; Stress; Survivorship; Breast Cancer; Dietary Habits
Keywords: breast cancer survivor; dietary omega-3 intervention; psychoneurological symptoms
MeSH Terms: conditions — Fatigue; Depression; Pain; Parasomnias; Breast Neoplasms; Feeding Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low Omega-3LC group (Experimental): Participants will consume a personalized meal plan for 2 weeks and consume an increased quantity of fish to 6 oz. wild salmon (1 steak, 6oz /steak)or 14.3 oz. (5.5 packs, 2.6 oz/pack) of chunk light tuna (1020 mg Omega-3LC/week) for 6 weeks.
  Interventions: Behavioral: Personalized Meal Plan; Behavioral: Dietary Omega-3LC intervention
- High Omega-3LC group (Experimental): Participants will consume a personalized meal plan for 2 weeks and consume an increased quantity of fish to 12 oz. wild salmon (2 steak,12 oz /steak)or 28.6 oz. (11 packs, 2.6 oz/pack) of chunk light tuna (2040 mg Omega-3LC/week) for 6 weeks.
  Interventions: Behavioral: Personalized Meal Plan; Behavioral: Dietary Omega-3LC intervention

INTERVENTIONS:
Behavioral: Personalized Meal Plan — Personalized dietary plans will be developed incorporating the NPAGCS, while personalizing the plan based upon anthropometric characteristics, gender, age and self-reported activity level upon entry into the investigation, goals, typical dietary consumption patterns, and food preferences. A trained research assistant will use the USDA MyPlate88 site (www.choosemyplate.gov) to enter participant characteristics and determine the appropriate calorie level. A daily checklist will be then generated outlining the number of daily servings that should be consumed for each food group. Information will also be provided regarding serving sizes for different foods in the respective food groups and education will be provided regarding tailoring personal dietary preferences to meet the guidelines. Participants will be provided with a printed copy of their meal plan and instructed to initiate it for a 8-week period.
Behavioral: Dietary Omega-3LC intervention — Following randomization, participants will be provided with fish to be consumed for 6 weeks. As a component of the dietary intervention, participants in high and low omega-3LC group will be provided with frozen, wild caught salmon (or if they dislike salmon, prepackaged, individual use foil packs of chunk light tuna). Salmon and chunk light tuna were chosen due to high omega-3LC content, low methylmercury content, low cost and ease of use. Vacuum packed, frozen salmon will be delivered to participants in large freezer bags and instructed to arrange visit times to ensure they can go directly home following the visit. Instructions for safe storage, fish handling and recipes to avoid fatigue of fish will be also be provided to participants when they receive the fish.

SUMMARY:
Inflammation has been consistently associated with psychoneurological symptoms (PNS) among breast cancer survivors (BCS). Evidence supporting interventional strategies promoting symptom-self management in reducing inflammation-induced PNS in BCS is limited. Current guidelines for BCS encourage the consumption of foods rich in omega-3 fatty acids. The omega-3 fatty acid docosahexaenoic acid (DHA), abundantly available in fish, has a role in inflammatory downregulation. Low dietary DHA has been associated with inflammation and fatigue in BCS. Dietary planning targeting increased fish consumption thereby reducing red and processed meats are components of the major nutritional recommendations for BCS. A critical gap exists in knowledge regarding interventions promoting adherence to dietary guidelines in BCS supporting PNS self-management. This investigation uses personalized meal planning among BCSs (n=150) who are 1-2 years post-treatment for early-stage breast cancer and experiencing PNS (pain, fatigue, depression, sleep disturbance, stress) to evaluate the feasibility of a personalized meal planning approach in supporting adherence to current dietary guidelines for BCS. As a first step in this program of research, we will evaluate the feasibility of an personalized meal planning approach in promoting adherence to dietary guidelines for BCS through evaluating the feasibility of a personalized meal planning approach in a cohort of BCSs with respect to recruitment, group allocation, salivary inflammatory quantification and receptivity to and adherence with dietary interventions. This investigation will also contribute to a preliminarily evaluation of the efficacy of high or low fish diet in reducing inflammation (IL-1β, IL-6, TNF-a) and PNS symptoms. Nationally, there is a priority for the development of personalized health strategies supporting self-management of adverse symptoms. This investigation focused on PNS in BCS is an initial step in generating new knowledge in efficacious approaches toward guiding decisions on dietary behavior change strategies that are personalized, cost-effective, and sustainable.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with BCA between 1 and 2 years prior to study enrollment
* completed chemotherapy (except tamoxifen/aromatase inhibitors) and/or radiation
* no evidence of cancer recurrence;
* no chronic medical conditions involving the immune system or regular use of immunosuppressive medications;
* no history of previous chemotherapy or cancer
* no diagnosis of dementia or active psychosis;
* 30-75 years of age
* Able/willing to sign informed consent.

Exclusion Criteria:

* Women not meeting the inclusion criteria above;
* Non English-speaking

Ages: 35 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2018-04-11 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline depressive symptom at week 10 | baseline, Week 3 and Week 10
  Epidemiological Studies Depression Scale is 20-item self-report instrument. Each item is scored 0-4 at a 4-point scale, yielding a total between 0 and 80. A higher score indicates a worse depressive symptom.
Change from baseline pain at week 10 | baseline, Week 3 and Week 10
  Brief Pain Inventory short form assesses the severity of pain, location of pain, pain medications, amount of pain relief in the past 24 hours or the past week, and the impact of pain on daily functions. Each item is scored 0-10 at a 10-point scale, with 0 representing no pain or no pain interference and 10 representing worst pain or complete pain interference. The mean of 4 severity items will be used as a measure of pain severity, and the mean of the 7 interference items will be used as a measure of pain interference.
Change from baseline fatigue at week 10 | baseline, Week 3 and Week 10
  Brief Fatigue Inventory short form is a 9-item scale to assess cancer-related fatigue and its impact on daily functioning. Each item score 0-10 at a 10-point scale. On the BFI, severe fatigue can be defined as a mean score of 7 or higher.
Change from baseline sleep disturbance at week 10 | baseline, Week 3 and Week 10
  The 21-item General Sleep Disturbance Scale consists of items evaluating various aspects of sleep disturbance (quality and quantity of sleep, sleep onset latency, number of awakenings, excessive daytime sleepiness, and medication use) over the past week. Items are rated on a scale ranging from 0 (never) to 7 (every day). All items are summed to produce a total score ranging from 0 (no sleep disturbance) to 147 (extreme sleep disturbance).
Change from baseline perceived stress at week 10 | baseline, Week 3 and Week 10
  Levels of stress will be measured by the 10-item Perceived Stress Scale. Each item is rated on a 5-point scale ranging from 0 (never) to 4 (very often). The final score is obtained by reversing responses to the four positively stated items and then summing across all scale items. A higher score represents a higher perceived stress.

SECONDARY OUTCOMES:
Change from baseline salivary inflammatory markers at week 10 | 3 years
  To quantify salivary inflammatory markers (CRP, IL-1β, IL-6, TNFα), salivary samples will be collected at baseline, week 3, and 10 during the study period. Salivary assay kits (multiplex) specific to the inflammatory markers of interest will be used to quantify salivary samples according to established protocols.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle P Judge, PhD, Principal Investigator — University of Connecticut
Locations (1):
- Hartford HealthCare Cancer Institue, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No